CLINICAL TRIAL: NCT02671370
Title: Cervical Range of Motion in Neck Pain Patients: A Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Swanenburg, Head of PT Research, Balgrist University Hospital
Other Study IDs: 2015-00049
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measurement of the range of motion of the cervical spine — There is no intervention. Only measurements and interviews are taken.

SUMMARY:
This study there are any associations between objective and subjective outcome measures, measuring the cervical range of motion and if the restriction matter to the patient.

DETAILED DESCRIPTION:
Objective and subjective outcome measures are frequently used assessments in clinical practice.

The investigators will use different subjective and objective outcome measures to evaluate any possible associations, as well as to investigate if restrictions of movement matters to patients.

Additionally to the assessments tools the investigators will use interviews to extend the scope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any duration of neck pain
* Men and women older than 18 years
* Signed informed consent

Exclusion Criteria:

* Disc herniation of the cervical spine
* Spinal canal stenosis
* Acute accidents
* Surgery of the cervical spine
* Pacemaker and / or defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with neck pain of any duration
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion (CROM) | Baseline
  The cervical range of motion will be measured using the CROM device

SECONDARY OUTCOMES:
Neck Disability Index | Baseline
  Questionnaire, measuring the subjective restriction of the participant during activities of daily living
S-ROM-Neck | Baseline
  Questionnaire, the participants will be asked to assess their ability to move there neck and if they feel restricted.
Interviews (personal,semi-structured guided, open-ended questions) in a one-to-one Setting. Recorded with a voice-recorder. | Baseline
  10 of the participants will be asked to also take part in an interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
no there is not